CLINICAL TRIAL: NCT04462887
Title: Developing Nursing Interventions to Enhance Recovery Following Sudden Cardiac Arrest
Brief Title: Nursing Interventions Following Sudden Cardiac Arrest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Cynthia M. Dougherty, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 13730; R01NR004766 (NIH)
Record Dates: First submitted 2020-06-16; First posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: ICD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nursing intervention program (Experimental): The nursing intervention program consisting of 3 parts: (1) Structural Informational (SI) booklet, (2) Nursing Telephone Support (NTS) protocol, and (3) Nurse Pager 24/7.
  Interventions: Behavioral: Nursing intervention program
- Usual Care Group (No Intervention): Usual care participants received treatment as usual from their health care providers.

INTERVENTIONS:
Behavioral: Nursing intervention program — The intervention consisted of structured information (SI) provided in a booklet, nursing telephone support (NTS) and access to a nurse pager 24h/day. The SI booklet, Sudden Cardiac Arrest: A Survivor's Experience, contains 2 components: a descriptive component including individual verbatim statements about experiences of others during the first year of recovery and a management component outlining successful strategies used by others in dealing with issues in recovery. The NTS telephone calls included: check-in about current concerns, assessment of the topic for the week, review of common recovery experiences, discussion of behavioral strategies for dealing with the topic for the week, provision of positive feedback for strategies already working well, anxiety reduction statements, practice of new behaviors using role-playing and problem solving techniques, summarization, setting specific goals for the upcoming week, and collaborating on a learning assignment for the subsequent week.
  Arms: Nursing intervention program

SUMMARY:
Determine the benefits of implantable cardioverter defibrillator (ICD) patients participating in a structured, 8-week educational telephone intervention delivered by expert cardiovascular nurses post-ICD. To determine if individuals participating in a post-hospital telephone nursing intervention would demonstrate (1) increased physical functioning, (2) increased psychological adjustment, (3) improved self-efficacy in managing the challenges of ICD recovery, and (4) lower levels of health care utilization over usual care at 1, 3, 6 and 12 months post-ICD implantation.

DETAILED DESCRIPTION:
The goal of the study was to determine if a short-term social cognitive theory intervention would improve physical functioning and enhance psychological adjustment after receiving a first time ICD. The central aim of this study was to determine if individuals participating in a telephone nursing intervention compared to usual care demonstrated (1) improved physical functioning, (2) improved psychological adjustment, 3) improved knowledge related to sudden cardiac arrest (SCA) and the ICD, and (4) lower levels of health care use over a 3-month period post-ICD.

ELIGIBILITY:
Inclusion Criteria:

* the ability to read, speak, and write English,
* having telephone access,
* willingness to be followed for 1 year.

Exclusion Criteria:

* significant clinical comorbidities that prevented their return home after hospitalization,
* younger than 21 years of age,
* Short BLESSED cognitive screening tool scores ≥10.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 1998-01-01 (Actual); Primary Completion 2003-12-31 (Actual); Study Completion 2003-12-31 (Actual)

PRIMARY OUTCOMES:
Patient Concerns Assessment (PCA) | Change in patient concerns from baseline to 12 months
  scores from 0 to 58 in which lower scores reflect fewer symptoms
SF-12 Short Form Health Survey (SF-12) | change in general health (SF-12) score from baseline to 12 months
  scores from 0 to 100 with higher scores representing better self-reported health
State-Trait Anxiety Inventory (STAI) | change in anxiety (STAI) score from baseline to 12 months
  Scores range from 20 to 80. Higher scores indicating greater anxiety.

SECONDARY OUTCOMES:
Number of ICD shocks | change in number of ICD shocks from baseline to 12 months
  The number of ICD shocks (if any) that the patient received from the ICD
Center for Epidemiologic Studies Depression Scale (CES-D) | change in depression (CES-D) score from baseline to 12 months
  Scores range from 0 to 60, with high scores indicating greater depressive symptoms.
Efficacy expectations: Sudden Cardiac Arrest Self Efficacy (SCA-SE scale) | change in efficacy expectations from baseline to 12 months
  SCA-SE scale has 2 sub-scales self-efficacy and self-management behavior. The first 8 items measure self-efficacy. Score for this sub-scale ranges from 0 to 8. higher the score greater is the self-efficacy.
Number of emergency room (ER) visits for ICD firings or cardiac arrhythmias | change in number of ER visits from baseline to 12 months
  The number of times a person went to the ER for evaluation over 12 months
Number of clinic visits related to the ICD | change in number of clinic visits from baseline to 12 months
  The number of times a person had an outpatient clinic visit for the ICD
Number of hospital admissions for ICD or cardiac related | change in number of hospital admission from baseline to 12 months
  The number of times a person stayed overnight, at least 24 hours, in the hospital.
Sudden Cardiac Arrest (SCA) Knowledge | change in SCA knowledge from baseline to 12 months
  Score ranges from 0 to 25. Higher the score greater is the ICD knowledge.
Heart rhythm stability | change in heart rhythm stability from baseline to 12 months
  self-reported number of cardiac arrhythmias and assessed using interrogation reports from ICD devices during routine follow-up visits
Self-management behavior: Sudden Cardiac Arrest Self Efficacy (SCA-SE scale) | change in self-management behavior from baseline to 12 months
  SCA-SE scale has 2 sub-scales self-efficacy and self-management behavior. The items - to 16 measure self-management behavior. Score range from 0 to 8 for self-management behavior skills. Higher the score greater is the self-management behavior skills.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia M. Dougherty, PhD, ARNP, Principal Investigator — University of Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dougherty CM, Johnson-Crowley NR, Lewis FM, Thompson EA. Theoretical development of nursing interventions for sudden cardiac arrest survivors using social cognitive theory. ANS Adv Nurs Sci. 2001 Sep;24(1):78-86. doi: 10.1097/00012272-200109000-00009. PMID 11554535
- [Result] Dougherty CM, Thompson EA, Lewis FM. Long-term outcomes of a telephone intervention after an ICD. Pacing Clin Electrophysiol. 2005 Nov;28(11):1157-67. doi: 10.1111/j.1540-8159.2005.09500.x. PMID 16359281
- [Result] Dougherty CM, Lewis FM, Thompson EA, Baer JD, Kim W. Short-term efficacy of a telephone intervention by expert nurses after an implantable cardioverter defibrillator. Pacing Clin Electrophysiol. 2004 Dec;27(12):1594-602. doi: 10.1111/j.1540-8159.2004.00691.x. PMID 15613121
- [Derived] Dougherty CM, Liberato ACS, Streur MM, Burr RL, Kwan KY, Zheng T, Auld JP, Thompson EA. Physical function, psychological adjustment, and self-efficacy following sudden cardiac arrest and an initial implantable cardioverter defibrillator (ICD) in a social cognitive theory intervention: secondary analysis of a randomized control trial. BMC Cardiovasc Disord. 2022 Aug 10;22(1):369. doi: 10.1186/s12872-022-02782-8. PMID 35948889